CLINICAL TRIAL: NCT06330454
Title: Multicenter Prospective Observational Study in Patients With Painful Total Knee Replacement and I-one Therapy
Brief Title: Painful Total Knee Replacement (TKA) and I-one Therapy
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Leo Massari, MD, University Hospital of Ferrara
Other Study IDs: 483/2020/Disp/AOUFe
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Knee Pain Swelling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Painfull TKA: Pulsed electromagnetic field therapy
  Interventions: Device: I-ONE

INTERVENTIONS:
Device: I-ONE — Pulsed Electromagnetic fields joint therapy

SUMMARY:
Arthroplasty operations are very frequent and their number is constantly increasing. The success of prosthetic surgery is linked to surgical factors (prosthesis type, prosthesis design, prosthesis material, surgical hand) and 'biological' factors (inflammation, pain, oedema, impingement). It is well known that important functional limitations may result mainly from an overreaction involving the peri-articular tissues. This is particularly true after total knee arthroplasty (TKA) surgery, during which a large part of the bone tissue and part of the peri-articular tissues (joint capsule, ligaments, synovium) are dislodged or removed. In the days following arthroplasty operations, the presence of a strong local inflammatory component is associated with pain and functional limitation, which usually resolves within a few months; however, it can sometimes take longer, and sometimes result in a chronic, albeit modest, inflammatory condition that lasts for years. There is still a percentage of 11-25% of patients who remain not completely satisfied with the result achieved with prosthetic surgery . Baker et al. state that 19.8% of patients experience pain one year after arthroplasty . Beswick et al. report that many patients (10-34%) continue to experience significant pain and functional limitation after arthroplasty even years later.

DETAILED DESCRIPTION:
The inflammatory response is mainly due to the presence of pro-inflammatory cytokines in the synovium; in fact, it has been shown that there is an inverse relationship between the amount of the pro-inflammatory cytokine IL-6 in the joint in patients undergoing TKA and the patient's functional recovery one month after surgery. It has also been shown that a high concentration in synovial fluid of catabolic factors, such as TNF-α, MMP-13 and IL-6, is predictive of a lower resolution of pain 2 years after prosthesis surgery. Sellam and Berenbaum emphasise the importance of considering the synovial membrane as a promising target for new therapeutic strategies to control inflammation and thus prevent joint problems or resolve clinical symptoms . There is an increasing need to find a local anti-inflammatory treatment to be implemented in the immediate post-surgery period to avoid chronic pain. Not only the pain condition, but also the functional condition, although better than the starting condition, cannot be considered completely satisfactory; 37% of patients one year after surgery have not achieved a complete functional recovery.

Extensive translational research has shown that biophysical stimulation with I-ONE® therapy (Pulsed Electromagnetic Field by IGEA SpA, Carpi, Italy) is able to modulate cartilage metabolism by increasing the reduction of the release of inflammation mediators involved in cartilage degeneration, such as inflammatory cytokines (IL-6 and IL-8) and lipid mediators of inflammation (prostaglandins E2), enhances the anti-inflammatory effect of individual adenosine agonists A2A and A3 by increasing the release of the anti-inflammatory cytokine IL-10.

In the clinic, I-ONE® therapy is able to prevent and/or slow down the degenerative phenomena that accompany surgery in patients with cartilage lesions treated with microfractures under arthroscopy in the knee or ankle, both in patients undergoing autologous chondrocyte transplantation in the presence of scaffolds at the knee , and in patients with osteochondral lesions of the talus, treated by graft transplantation, with addition of bone marrow concentrate. I-ONE® therapy has also proven effective in patients undergoing total knee replacement with or without patella prosthesis and after reverse shoulder replacement surgery.

Postoperative noninvasive therapy with the use of PEMF in patients with painful TKA resulted in significant improvement in pain and functional recovery, as demonstrated by the preliminary results of this prospective cohort study.

The study plans to recruit patients with painful TKA whose pain occurred from at least 30 days after surgery to a maximum of 180 days after surgery. All patients will be instructed to use local non invasive biophysical therapy with I-ONE® therapy (1.5 mT, 75 Hz) for 4 hours a day for 60 days. Clinical evaluations such as Visual Analog Score (VAS), SF-12 Health Survey (SF-12), EuroQol (EQ-5D) are scheduled at 1 month, 2, 6, 12 and 24 months after PEMF treatment; Knee Society Score (KSS) is scheduled at 3 months of follow-up. The use of nonsteroidal anti-inflammatory drugs (NSAIDs) is also recorded. Patients will be analyzed into three different groups based on the time elapsed between surgery and the beginning of PEMF therapy: Group 1 (30-90 days), Group 2 (91-150 days) and Group 3 (151-180 days).

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* painful total knee replacement at least 30 ± 3 days post-op up to a maximum of 180 ± 3 days post-op
* VAS ≥ 5
* absence of infection

Exclusion Criteria:

* pain caused by mechanical problems (misalignment, mobilisation, etc.),
* the presence of hip prostheses,
* previous knee infections,
* rheumatoid arthritis
* autoimmune diseases
* systemic diseases
* tumours
* major axial deviations
* obesity (BMI > 30 kg/m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients, orthopaedic clinic
Sampling Method: Probability Sample
Enrollment: 237 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2025-10-21 (Estimated); Study Completion 2025-10-21 (Estimated)

PRIMARY OUTCOMES:
Evaluate pain resolution after treatment with I-ONE® therapy in patients with painful TKA at least 1 month after surgery. | baseline, 30 days, 60 days, 180 days, 1 year, 2 years
  Visual analogue scales (VAS, 0 is the minimum and 10 is maximum values) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid classification of symptom severity and disease control.

SECONDARY OUTCOMES:
reduced NSAID intake | baseline, 30 days, 60 days, 180 days, 1 year, 2 years
  NSAID usage registration
improved recovery of joint function | baseline, 30 days, 60 days, 180 days, 1 year, 2 years
  The SF-12 (12-Item Short Form Surveyis range from 0 to 100) a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.

CONTACTS AND LOCATIONS:
Overall Officials: Leo Massari, MD, Principal Investigator — Azienda Ospedaliera-Universitaria Arcispedale S. Anna di Ferrara
Locations (7):
- Italy (7):
  - IRCCS Istituto Ortopedico Rizzoli, Bologna, BO
  - Poliambulanza Brescia, Brescia, BS
  - Policlinico San Matteo Pavia, Pavia, PV
  - Ospedale Mauriziano Torino, Torino, TO
  - Ospedale Sacro Cuore Don Calabria Negrar Verona, Negrar, VR
  - Policlinico di Bari, Bari
  - Ospedale Santo Spirito in Sassia/Ospedale San Filippo Neri Roma, Roma

IPD SHARING:
Plan to Share IPD: Undecided